CLINICAL TRIAL: NCT01564381
Title: Effects of Resveratrol Supplements on Vascular Health in Postmenopausal Women
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Gateway Health Alliance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 270881
Record Dates: First submitted 2012-02-22; First posted 2012-03-27 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Resveratrol (Experimental): The capsules will contain 90mg of resveratrol.
  Interventions: Dietary Supplement: Resveratrol
- ResA (Experimental): ResA is a product produced by using patented technology that physically binds resveratrol to arginine, creating a novel conjugate. The capsules will contain 90mg of resveratrol.
  Interventions: Dietary Supplement: ResA
- Placebo (Placebo Comparator): The placebo will be cellulose.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: ResA — 90mg of resveratrol conjugated with arginine.
  Arms: ResA
Dietary Supplement: Resveratrol — 90mg of resveratrol.
  Arms: Resveratrol
Dietary Supplement: Placebo — Made up of cellulose.
  Arms: Placebo

SUMMARY:
The investigators hope to learn if resveratrol supplementation can be beneficial for the cardiovascular system. Seeing that resveratrol is rapidly metabolized, the investigators are interested in learning if a novel form of resveratrol, ResA, which is a mixture of resveratrol with amino acid, may have greater bioavailability and lead to greater improvement in vascular function, compared to standard resveratrol supplement.

DETAILED DESCRIPTION:
Cardiovascular disease is the leading cause of morbidity and mortality in the United States. To reduce the risk of cardiovascular disease (CVD) and its associated health care costs, nutrition and health recommendations strongly advocate the consumption of a diet rich in fruits and vegetables. In addition to essential vitamins and minerals, fruits and vegetables contain a number of bioactive compounds that may be involved in vascular function.

The "French Paradox" refers to diet patterns that, despite being high in saturated fat, are associated with a relatively low cardiovascular risk. An important aspect of many of the diets that were identified in the French Paradox studies is a significant intake of wine, particularly red wine, which can contain an array of phytochemicals that have been postulated to improve cardiovascular health. A polyphenolic that has received particular attention is this regard is resveratrol.

The stilbene resveratrol is found predominately in red grapes, red wine, peanuts and some berries, and it has been touted in the popular press for its potential health-promoting benefits. Emerging evidence suggests a role for resveratrol in the protection against numerous degenerative health problems including CVD and certain cancers, diabetes and some forms of neurodegeneration.

The amount of resveratrol in most foods is very low; thus obtaining the amounts of this compound that have been associated with improved health in animal models is difficult for humans. ResA is a product produced using patented technology that physically binds resveratrol to arginine, creating a novel conjugate. In the preliminary studies the ResA conjugate produced higher peak plasma levels, as well as total plasma levels that persist for a longer period of time when fed to rats. Whether similar results would occur in humans, and the extent to which increasing blood resveratrol concentration can be associated with positive cardiovascular effects in an at-risk population is the subject of this project.

ELIGIBILITY:
Inclusion Criteria:

* 50 to 70 years of age
* Lack of menses in the last year and FSH 23-116.3 mlU/mL
* Subject is willing and able to comply with the study protocols.
* Subject is willing to consume resveratrol supplements/placebo capsules on three separate occasions.
* BMI 18.5-34.9 kg/m2
* Weight ≥ 110 pounds
* LDL-C ≥ 130 mg/dL

Exclusion Criteria:

* BMI ≥ 35 kg/m2
* Self reported use of anticoagulation agents including NSAIDs
* Self reported use of oral cortisone or other immunosuppressive agents,
* Self reported underlying neoplasia or immunological disease
* Food faddists or those taking a non-traditional diet
* Self reported physical activity restricted or reduced due to chronic health conditions
* Self reported diabetes
* Blood pressure ≥ 140/90 mm Hg
* PFA-100 readings 10 % outside of normal reference range (normal reference range for ADP-Collagen: 71-118 sec; Epinephrine-Collagen: 94-193 sec).
* Self reported renal or liver disease
* Self reported heart disease, which includes cardiovascular events and stroke
* Self reported Cushing's syndrome
* Self reported chronic/routine high intensity exercise
* Inability to properly place or wear the PAT probes or abnormal measurements on pre-screening PAT
* Abnormal Liver, CBC or Chemistry panels (laboratory values outside the reference range) if determined to be clinically significant.
* Self reported cancer within past 5 years
* Self reported history of psychiatric disorders i.e. schizophrenia or bi-polar or depression treated with antidepressants within the last 1 year.
* Self reported use of MAOI inhibitor within the last 1 year (e.g. phenelzine (Nardil), tranylcypromine (Parnate), etc)
* Self reported malabsorption (e.g. difficulty digesting or absorbing nutrients from food,

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Bioavailability of a novel formulation of resveratrol (ResA) compared to a standard resveratrol supplement | up to 2 hour after consumption
  We will assess metabolites concentrations of resveratrol and ResA in plasma via HPLC method.
Change in vascular function in response to ResA compared to native resveratrol | up to 2 hours after consumption
  We will assess changes in vascular function measured by peripheral arterial tonometry.

SECONDARY OUTCOMES:
Change in platelet reactivity in response to ResA intake | 1 hour after consumption
  We will assess platelet function in response to ADP, collagen and arachidonic acid as measured by platelet aggregometer.

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Hackman, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis - Ragle Human Nutrition Research Center, Davis, California, United States